CLINICAL TRIAL: NCT00526279
Title: A Prospective, Non-interventional, Observational, Multi-center Trial to Evaluate Compliance and Efficacy in Mono and Combination Treatment of Candesartan Cilexetil(Atacand)/ Candesartan Cilexetil 16mg, Hydrochlorothiazide 12.5mg(Atacand Plus) in Hypertension
Brief Title: COmpliance and Efficacy in Mono and Combination Tablet Study ATacand/Atacand Plus
Acronym: COMBAT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-CKR-ATA-2007/2
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Hypertension
Keywords: Hypertension; Atacand/Atacand plus; COMBAT; Compliance; Naturalistic; Observational
MeSH Terms: conditions — Hypertension; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate compliance and patients' satisfaction in mono and combination treatment of Candesartan cilexetil (Atacand)/ Candesartan cilexetil 16mg, hydrochlorothiazide 12.5mg (Atacand plus) in hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have consented to participation/data release in this study
2. Patients diagnosed with hypertension and prescribed with atacand/atacand plus by the physician based on clinical decision

Exclusion Criteria:

1. Secondary hypertension requiring therapy other than antihypertensive medication
2. Patients not prescribed with atacand/atacand plus based on safety reasons or any other reason as determined by the physician
3. Women in pregnancy or lactation
4. Patients enrolled in any other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care
Sampling Method: Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyunah Caroline Choi, Study Director — AstraZeneca Korea
Locations (3):
- South Korea (3):
  - Research Site, Seoul, Jongro-gu
  - Research Site, Seoul, Kangnam-gu
  - Research Site, Seoul, Songpa-gu